CLINICAL TRIAL: NCT02786914
Title: Nut Cross-Reactivity - ACuiring Knowledge for Elimination Recommendations (NUT-CRACKER) Study
Brief Title: Predictors of Positive Food Challenge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 235/14
Record Dates: First submitted 2016-05-05; First posted 2016-06-01 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Oral Immunotherapy for Food Allergy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with suspected tree-nut or sesame allergy based on sensitization on skin-prick tests (SPT), will be assessed for allergy using component analysis and basophil activation test (BAT) and entered into oral immunotherapy (OIT). Component analysis and BAT will be repeated after completion of OIT. Patients with tree-nut or sesame allergy treated with the standard of care of elimination diet will serve as controls

DETAILED DESCRIPTION:
Patients will be recruited from the pool of patients referred to the investigators center for evaluation of food allergy. For each tree-nut (walnut, pecan, cashew, pistachio, hazelnut or almond) evaluated, 30 patients (ages 4-45 years old), with allergy to at least one tree-nut will be recruited from the database pool referred to above. Skin prick tests (SPT) using standardized 10 mg/ml tree-nut extracts, and BAT will be performed for all suspected allergens. Sera will be taken and sent to ThermoFisher for IgE and IgG4 binding analysis to purified components. Open OFCs will be performed for each tree-nut, unless clinically contraindicated. The results of the OFC will form the basis to determine the sensitivity and specificity of the component testing. Similarly, 40 patients with suspected sesame allergy will be administered SPT and component analysis for sesame, with correlations to OFC.

The investigators will also utilize BAT to directly test whether the identified purified components are sufficient to elicit reactivity. This objective can be met by either utilizing saved patient sera on naive basophils or directly on a subsequently obtained blood sample from the patient. For patients enrolling in OIT (secondary objective), sera will also be taken after completion of the therapeutic regimen, and IgE as well as IgG4 binding to the same components will be assessed and compared to pre-OIT results.

4.2 STATISTICAL ANALYSIS AND METHODS

4.3 Patients will be grouped by OFC their allergy status result for each tree-nut (patients with a documented IgE-mediated reaction in the previous year or a positive OFC vs. patients with regular consumption of the index food or a negative OFC). Descriptive statistics (proportions for categorical variables, means or medians and standard deviations or inter-quartile range for continuous variables) will be reported for all key participant variables, including baseline and demographic characteristics, SPT, BAT and component testing results.

For the primary objective, the sensitivity and specificity of the diagnostic tests (wheal for SPT, and CD63 induction for BAT) and IgE/IgG4 binding to the purified components in predicting OFC results allergy will be compared by receiver operating characteristic (ROC) analysis. To this end, the investigators will evaluate molecular allergens singly or in groups for their predictive utilities.

For the secondary objective, OFC positive patients with documented allergy who undergo OIT for tree-nuts (n=15 for each tree-nut) or sesame (n=15) will be grouped according to OIT outcome. Paired t-tests comparing IgE and IgG4 binding of specific molecular allergens in individual patients before and after treatment will be performed. Additionally, the pre-OIT IgE and IgG4 profiles against particular molecular allergens will be compared between OIT outcome groups by t-test. 10 control patients treated with the standard of care of elimination diet will be compared.

Power analysis: Using the Pearson Chi-square test for two proportions, with the assumption that 75% of all OFC+ to tree-nuts will be positive to at least one specific component, in order to detect a result with a P-value of <0.05, 15 positive and 15 negative sera for each tree-nut would yield a power of 0.816. Based on the investigators experience with immunoreactivity as assessed by western blot, in fact the investigators would expect that much more than 75% of OFC+ patients would show IgE reactivity against at least one component. Thus, the investigators feel that a total of thirty sera for each tree-nut should suffice for the analysis.

Total number of patients: 180 patients to be evaluated for tree-nut allergy and 40 for sesame allergy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4-45 years old, with a positive SPT to tree-nuts (walnut, pecan, cashew, pistachio, hazelnut or almond) and/or sesame, and either a history of a reaction in the past year, a positive OFC, or patients refraining from tree-nut consumption.

Exclusion Criteria:

* A history of other numerous chronic inflammatory diseases, including inflammatory bowel disease and other autoimmune diseases.

Ages: 4 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be recruited from the pool of patients referred to our center for evaluation of food allergy. The investigators have a database of over 1200 food allergic patients (OFC+) that can be utilized to attain the recruitment goal.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive food challenge to tree-nuts and sesame | 1 year
  Determining the best diagnostic method that would predict a positive vs. negative oral food challenge in food sensitized patients

SECONDARY OUTCOMES:
Number of patients with decreased component reactivity for a particular tree-nut and for sesame following OIT | 2.5 years
  To determine how many patients have decreased reactivity following successful desensitization to the same food in OIT
Number of patients with decreased component cross reactivity for a particular tree-nut and for sesame following OIT | 2.5 years
  To determine how many patients have decreased component reactivity following successful desensitization to a different food in OIT

CONTACTS AND LOCATIONS:
Locations (1):
- The institute of Allergy, Immunology and Pediatric Pulmonary Medicine, Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No